CLINICAL TRIAL: NCT06663046
Title: A Clinical Study Evaluating the Safety and Efficacy of Universal BCMA-Targeted CAR-T (UWD-00B) Therapy for Refractory and Relapsed Multiple Myeloma
Brief Title: Universal CAR-T Cells (REVO-UWD-00B) for Refractory and Relapsed Multiple Myeloma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wondercel Biotech (ShenZhen) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-REVO-UWD-BCMA
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myleoma; Refractory and Relapsed Multiple Myeloma
Keywords: BCMA; REVO-U platform; Off-the-shelf CAR-T therapy
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Off-the-shelf REVO-UWD-00B (Experimental): Eligible participants will undergo FC lymphodepleting chemotherapy preconditioning, followed by a one-time injection of universal UWD-00B cells
  Interventions: Biological: Single dose injection of certain dose of UWD-00B; Drug: MMF Immunosuppression

INTERVENTIONS:
Biological: Single dose injection of certain dose of UWD-00B — Eligible participants will undergo FC lymphodepleting chemotherapy preconditioning after signing an informed consent form, followed by a one-time injection of certain dose of universal UWD-00B cells
Drug: MMF Immunosuppression — One day after the completion of fludarabine preconditioning (D-2), initiate oral mycophenolate sodium at a dose of 1440 mg twice daily (BID) for 15 consecutive days, or extend the duration appropriately based on CAR-T cell expansion status (discontinuation may occur at the end of CAR-T cell expansion or on the day of patient discharge). The maximum duration of administration must not exceed 30 days.

SUMMARY:
This study is a single-arm, investigator-initiated clinical trial. The primary objective is to evaluate the safety and preliminary efficacy of administering universal BCMA CAR-T cells to subjects with refractory and relapsed multiple myeloma. Eligible participants will undergo FC preconditioning after signing an informed consent form, followed by a one-time injection of universal UWD-00B cells to assess its safety and efficacy. Subjects will be hospitalized for a period, and after discharge, they will undergo periodic efficacy assessments and long-term survival follow-up for at least five years.

DETAILED DESCRIPTION:
Multiple myeloma is a malignant plasma cell disease with high mortality rates. Patients with relapsed and refractory cases, especially those resistant to conventional therapies (immunomodulators, proteasome inhibitors, and anti-CD38 monoclonal antibodies), typically have limited survival. CAR-T cell therapy is a cutting-edge approach in which T cells are genetically modified to target cancer cells. UWD-00B is designed to target BCMA, a protein highly expressed on myeloma cells but minimally present in other body tissues, making it an ideal target. Previous BCMA CAR-T therapies have shown promise, but production limitations make universal, off-the-shelf products like UWD-00B critical for broader patient accessibility.

Primary Objective is to evaluate the safety and initial efficacy of UWD-00B in patients with r/r MM. The secondary Objectives is to investigate pharmacokinetic (PK) and pharmacodynamic (PD) characteristics, including the persistence and effectiveness of UWD-00B in targeting BCMA-positive cells. This study will enroll approximately 30 patients with relapsed or refractory MM, aged 18-75. Following preconditioning chemotherapy to enhance CAR-T cell efficacy, patients will receive a single infusion of UWD-00B. The study spans multiple phases, including screening, infusion, and a two-year follow-up to assess both short- and long-term safety and efficacy.

This study hopes to provide data supporting UWD-00B as an effective, accessible treatment for r/r MM, potentially paving the way for similar universal CAR-T therapies in other cancers.

ELIGIBILITY:
Inclusion Criteria:

* The patient or their guardian understands and voluntarily signs the informed consent form and is expected to complete the study's follow-up assessments and treatments.

Age between 18 and 75 years, with no gender restrictions. Diagnosis of multiple myeloma according to the International Myeloma Working Group (IMWG) criteria.

Documented evidence of relapsed/refractory or primary refractory multiple myeloma, defined as follows:

Relapsed/Refractory: Lack of response to salvage therapy (defined as no minimal response (MR) or disease progression during treatment), or disease progression within 60 days of the last treatment, or progression after achieving MR or better.

Primary Refractory: No response (MR or better) to any previous treatment, with no clinical progression or minimal M-protein change, or meeting criteria for primary refractory progression.

Presence of measurable disease at screening by any of the following criteria: serum M-protein ≥ 1.0 g/dL, urine M-protein ≥ 200 mg/24 hours, or for light-chain myeloma without measurable disease in serum or urine, serum free light chain (FLC) ≥ 10 mg/dL with abnormal serum immunoglobulin κ/λ FLC ratio.

Resolution of prior treatment-related toxicities to Grade <2 per CTCAE (unless related to underlying malignancy or deemed stable and not impacting safety or efficacy).

ECOG performance status 0-2 and an expected survival of more than 3 months.

Laboratory values meeting the following standards, indicating adequate organ and marrow function, with no severe hematological or organ impairment:

Serum albumin ≥ 25 g/L Hemoglobin ≥ 8.0 g/dL (without RBC transfusion in the prior 7 days; recombinant human erythropoietin permitted) Absolute neutrophil count ≥ 0.75×10⁹/L (growth factor support allowed if discontinued ≥7 days before test) Platelet count ≥ 60×10⁹/L (no platelet transfusion within 7 days) Creatinine clearance ≥ 30 mL/min/1.73 m² (using kidney disease formula or 24-hour urine collection) ALT and AST ≤ 3.0×ULN Total bilirubin ≤ 2.0×ULN (Gilbert's syndrome exception with direct bilirubin ≤ 1.5×ULN) PT and APTT < 2×ULN Blood oxygen saturation ≥ 95%

Exclusion Criteria:

* Diagnosis or treatment of other invasive malignancies within 3 years, with the exception of curatively treated non-melanoma skin cancer or malignancies with no active disease for ≥ 3 years.

Prior anti-cancer treatments within 14 days or 5 half-lives (whichever is shorter) including targeted therapy, epigenetic therapy, or investigational drugs, monoclonal antibody therapy within 21 days, proteasome inhibitor therapy within 14 days, immunomodulators within 7 days, or radiotherapy (except if the radiotherapy field covers ≤5% of bone marrow).

Known active CNS involvement or clinical evidence of myelomatous meningitis. Diagnosis of Waldenström macroglobulinemia, POEMS syndrome, or primary AL amyloidosis at screening.

Positive for HBsAg or HBcAb with HBV DNA >1000 copies/mL; positive for HCV antibodies, HIV antibodies, CMV DNA, syphilis, or EBV DNA.

History of severe allergies, including anaphylaxis, or known allergy to any study drugs, their components, or murine proteins.

Serious cardiac conditions, including but not limited to severe arrhythmias, unstable angina, recent myocardial infarction (within 6 months), NYHA Class III/IV heart failure, recent CABG, unexplained syncope, severe non-ischemic cardiomyopathy, or uncontrolled hypertension.

Unstable systemic diseases deemed significant by the investigator, including severe liver, renal, or metabolic disorders.

History of acute or chronic graft-versus-host disease (GVHD) or currently on immunosuppressive therapy for GVHD within 6 months prior to screening.

Active autoimmune or inflammatory neurologic diseases such as Guillain-Barré syndrome, ALS, or clinically significant cerebrovascular diseases.

Presence of urgent tumor-related emergencies requiring immediate treatment, such as spinal cord compression, bowel obstruction, leukostasis, or tumor lysis syndrome.

Uncontrolled bacterial, fungal, viral, or other infections requiring antibiotics.

Major surgery within 4 weeks prior to lymphodepletion, or planned major surgery during the study period.

Live virus vaccinations within 4 weeks prior to screening. Severe psychiatric illness. History of alcohol or substance abuse. Pregnant or lactating women, or females and males planning to conceive within 2 years post-cell infusion.

Any contraindication to study procedures or conditions deemed by the investigator to pose an unacceptable risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Within the first month post-infusion.
  The highest dose of UWD-19 CAR-T cells that can be administered without causing unacceptable side effects, measured during the dose escalation phase.
Dose-Limiting Toxicities (DLT) | Within the first month post-infusion.
  The incidence of treatment-related toxicities that prevent further dose escalation.
Treatment-Emergent Adverse Events (TEAE) | From the administration of UWD-00B CAR-T cells through six months post-infusion
  The frequency and severity of adverse events that arise following the administration of UWD-00B CAR-T cells.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Measured at 3 and 6 months after treatment
  The proportion of patients with a measurable efficacy (complete or partial response) following UWD-00B CAR-T therapy.
Progression-Free Survival (PFS) | From the start of treatment up to 5 years
  The length of time during and after treatment that the patient lives without disease progression.
Overall Survival (OS) | From the start of treatment up to maximum follow-up period of five years
  The duration from the start of treatment to the time of death from any cause.
Duration of Response (DOR) | From the administration of UWD-00B CAR-T cells to a maximum follow-up period of five years
  The time from initial response (CR or PR) to disease progression or relapse or any cause of death.

CONTACTS AND LOCATIONS:
Overall Officials: Pengcheng He, M.D. Ph.D., Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No